CLINICAL TRIAL: NCT07053826
Title: Prospective, Randomized, Controlled Trial to Evaluate the Effect of Preoperative Penile Traction Therapy on Post-penile Implant Length and Patient Satisfaction
Brief Title: Penile Lengthening Pre-Penile Prosthesis Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pathright Medical (Unknown)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Professor and Endowed Chair of Plastic Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24110037
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Inflatable Penile Prosthesis; Penile Traction Therapy; RestoreX; Penile Enlargement
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a double-armed, controlled, open-label randomized trial assessing the above outcomes in the presence or absence of preoperative penile traction device (RestoreX) use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Penile Prosthesis Implantation (Active Comparator): Patients with erectile dysfunction presenting for placement of a three-piece inflatable prosthesis who are randomized to the no intervention arm will proceed directly to implantation of a standard-of-care inflatable penile prosthesis at the next available surgical appointment. They will not use the RestoreX penile traction device. They will complete standardized assessments of sexual function and satisfaction before and after placement.
  Interventions: Procedure: Inflatable Penile Prosthesis Implantation
- RestoreX and Penile Prosthesis Implantation (Experimental): Patients with erectile dysfunction presenting for placement of a three-piece inflatable prosthesis who are randomized to the intervention arm will be provided with a RestoreX penile traction device, which they will utilize for three months prior to implantation of a standard-of-care inflatable penile prosthesis. They will complete standardized assessments of sexual function and satisfaction before and after placement, as well as a device use diary.
  Interventions: Device: Penile Traction Device; Procedure: Inflatable Penile Prosthesis Implantation

INTERVENTIONS:
Device: Penile Traction Device — Patients will be randomized into one of two groups: penile traction therapy 30 min 3x/day x 3 months, or control (no treatment). Preoperative erectile function surveys will be recorded in the EMR per standard of care. Following randomization, patients allocated to the treatment arm will be instructed how to use the device properly. Patients in the treatment arm will record a daily journal of use of the device (Appendix 1). After a minimum of 3 months, patients in the treatment arm will return for their scheduled procedure. Control arm patients will be scheduled directly for an OR date.
  Other Names: RestoreX; PTT
  Arms: RestoreX and Penile Prosthesis Implantation
Procedure: Inflatable Penile Prosthesis Implantation — Implantation of a three-component inflatable penile prosthesis.

SUMMARY:
The goal of this study is to determine whether or not the use of a penile traction therapy device known as RestoreX prior to implantation of a penile prosthesis can increase the length of the implant used during surgery. The device used in this study is commercially available and has been used successfully to facilitate penile lengthening in patients with diabetes and after a certain type of prostate surgery. Use of the device has not been shown to have any detrimental effects on sexual or overall health.

DETAILED DESCRIPTION:
Men with erectile dysfunction (ED) refractory to medical therapies are often recommended to undergo placement of an inflatable penile prosthesis (IPP). However, men commonly report a perceived loss of penile length following IPP implantation. This is likely due to one of several factors, including the underlying disease process which resulted in loss of penile length, effects of aging on penile length (loss of elasticity; increased fibrosis), changes in abdominal physiology (development of pre-pubic fat pad that obscures the penis), and recall bias (incorrect recollection of prior penile length).

Several attempts have been made by investigators to optimize penile length prior to placement of the penile prosthesis, including adjunctive surgical maneuvers (excision of suprapubic fat pad, release of suspensory ligament, direct penile extension), use of injectable materials, and pre-operative use of penile traction therapy (PTT). In a small pilot study of 10 men undergoing IPP, Levine and colleagues recommended the use of the Andropenis PTT ≥2 hrs daily for 2-4 months. At 15 months follow-up, patients achieved a +1.6 cm increase compared to pre-traction stretched length, and +0.9 cm increase following prosthesis implantation. Results from a non-validated satisfaction questionnaire demonstrated that no patients reported loss of length following surgery. Unfortunately, the study did not include a control group, thus limiting the conclusions which may be drawn.

Compared to other options, PTT offers several potential advantages in that it is minimally invasive, does not increase the morbidity of surgery, and has not been shown to result in any long-term side effects. RestoreX is a commercially available PTT device that was developed by the Mayo clinic and has been licensed to PathRight Medical. It has been designated as a Class I device that does not require clinical human trials. The device is currently utilized in 30-minute intervals, with up to 3 sessions performed per day, and has demonstrated efficacy at increasing stretched penile length in patients with postprostatectomy penile shortening and diabetes mellitus.

Given the clinical issue of dissatisfaction with penile length post IPP, the potential role for PTT, and the limited amount of data that are currently available, we seek to perform a clinical trial evaluating the effect of PTT stretched penile length, size of prosthetic implantation at time of surgery, and patient satisfaction following implantation.

The device has two functional aspects. The first is the ability to provide direct traction on the penis. The second is the ability to provide counter-bending forces, to treat conditions such as Peyronie's disease. In the current study, only the direct traction aspects of the device will be investigated. Men randomized to treatment will be recommended to utilize the device for 30 minutes, 3 times daily for 3 months prior to placement of an IPP, with up to 1.3 additional months to account for variability in surgical timing.

To date, the efficacy of the RestoreX device has been studied in multiple clinical trials, the results of which are briefly outlined below:

* In a randomized, controlled clinical trial, 82 men who underwent prostatectomy for prostate cancer revealed an average increase in stretched penile length of 1.6 cm after 5 months of RestoreX use vs no change for controls (P=0.001). Adverse events were transient and mild, with 87% of men reporting a desire to repeat therapy and 93% of participants reporting that they would recommend it to others.
* In the open-label phase of the study, the benefits of therapy were found to be maintained even after therapy was discontinued.
* In a randomized, single-blind, controlled trial, 110 men with Peyronie's disease were assigned 3:1 to penile traction therapy for three months vs no therapy. At three months, penile traction therapy was associated with a 1.5 cm increase in penile length and 11.7 degree reduction in penile curvature relative to controls. Further, erectile function scores improved 4.3 points relative to a loss of 0.7 points in the control group. The therapy was well tolerated; adverse events were transient and mild.
* Preliminary data also suggest that the RestoreX device can increase penile length on men with diabetes who did not undergo surgery.

Very limited data are available on the efficacy of PTT in men undergoing placement of an IPP. As noted above, a small pilot study of 10 men undergoing IPP demonstrated a +1.6 cm increase in penile length compared to pre-traction stretched length and 0% of men reporting loss of length following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of erectile dysfunction
* Can provide informed consent
* Are willing and able to comply with study procedures and visit schedules
* Are to be scheduled for a planned standard of care implantation of an inflatable penile prosthesis

Exclusion Criteria:

* Prior ischemic priapism
* Prior implantation of a penile prosthesis
* Prior use of any penile traction device
* Any prior penile surgeries other than circumcision
* Prior pelvic radiation
* Current or prior androgen deprivation therapy
* Active genital infection
* History of neophallus creation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Penile Length | At screening to approximately three months after enrollment at the time of penile prosthesis implantation
  Change in stretched penile length measured at time of enrollment and intraoperatively at the time of IPP implantation, measured in cm.
Prosthesis size | 0-4 months after enrollment at the time of penile prosthesis implantation
  Size of inflatable penile prosthesis cylinders placed
Sexual Satisfaction | At enrollment and at three-month postoperative follow up.
  Change in patient-reported satisfaction with their sexual function from enrollment to final postoperative follow up using the validated IIEF-15 (International Index of Erectile function - 15 item) questionnaire, which has a minimum score of 6 and maximum score of 75 with a larger number indicating improved sexual satisfaction. The change seen in participants assigned to the RestoreX device arm will be compared to the change seen in patients assigned to the control arm.
Incidence of Satisfaction with Penile Length | 3-8 months postoperatively
  A comparison of the incidence of participants reporting satisfaction with their penile length, expressed as a percentage or all participants within each group, based on participant reporting to an investigator during their surgical follow up.

SECONDARY OUTCOMES:
Compliance with Therapy | 0-4 months after enrollment, intervention arm only
  Patient compliance with traction device regimen using a device use diary will be assessed. Compliance will be reported as a percentage of recommended use sessions completed.
Incidence of adverse events | 0-16 months
  The incidence of all adverse events arising from penile traction therapy device use or inflatable penile prosthesis placement will be monitored throughout the study during in-person encounters and via chart review at the conclusion of the study.
Patient Satisfaction with Prosthesis Use | 3-7 months
  Patient satisfaction with their penile prosthesis will be assessed postoperatively using the validated Quality of Life and Sexuality after Penile Prosthesis (QoLSPP) survey, a 16-item survey with a maximum score of 80 and minimum score of 0, where a higher score corresponds to increased satisfaction. Scores of patients undergoing prosthesis placement alone will be compared to those of patients undergoing RestoreX therapy prior to prosthesis placement.
Patient Satisfaction with Prosthesis Use | 3-8 months
  Patients randomized to RestoreX device use prior to prosthesis placement will be asked if they would use a penile traction device again, and how satisfied they were, on surveys administered immediately prior to, and three months following, prosthesis placement using Likert-style questions.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Mercy Hospital, Urology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of the patients involved in the study, we do not plan to share IDP.

REFERENCES:
- [Background] Ziegelmann M, Savage J, Toussi A, Alom M, Yang D, Kohler T, Trost L. Outcomes of a Novel Penile Traction Device in Men with Peyronie's Disease: A Randomized, Single-Blind, Controlled Trial. J Urol. 2019 Sep;202(3):599-610. doi: 10.1097/JU.0000000000000245. Epub 2019 Aug 8. PMID 30916626
- [Background] Zganjar A, Toussi A, Ziegelmann M, Frank I, Boorjian SA, Tollefson M, Kohler T, Trost L. Efficacy of RestoreX after prostatectomy: open-label phase of a randomized controlled trial. BJU Int. 2023 Aug;132(2):217-226. doi: 10.1111/bju.16033. Epub 2023 May 9. PMID 37088866
- [Background] Toussi A, Ziegelmann M, Yang D, Manka M, Frank I, Boorjian SA, Tollefson M, Kohler T, Trost L. Efficacy of a Novel Penile Traction Device in Improving Penile Length and Erectile Function Post Prostatectomy: Results from a Single-Center Randomized, Controlled Trial. J Urol. 2021 Aug;206(2):416-426. doi: 10.1097/JU.0000000000001792. Epub 2021 Jun 1. PMID 34060339
- [Background] Trost LW, Munarriz R, Wang R, Morey A, Levine L. External Mechanical Devices and Vascular Surgery for Erectile Dysfunction. J Sex Med. 2016 Nov;13(11):1579-1617. doi: 10.1016/j.jsxm.2016.09.008. PMID 27770853
- [Background] Levine LA, Rybak J. Traction therapy for men with shortened penis prior to penile prosthesis implantation: a pilot study. J Sex Med. 2011 Jul;8(7):2112-7. doi: 10.1111/j.1743-6109.2011.02285.x. Epub 2011 Apr 14. PMID 21492409